CLINICAL TRIAL: NCT04875312
Title: Effect of Ultrasound Cavitation Versus Electro Acupuncture on Sex Hormones in Obese Infertile Patients With Polycystic Ovarian Syndrome
Brief Title: Effect of UC Versus EA on Sex Hormones in Obese Infertile Patients With PCOs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohamed Abdel Hamid elgaedy (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abdel Hamid elgaedy, Head OF physical therapy in AGA hospital, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003187
Record Dates: First submitted 2021-04-19; First posted 2021-05-06 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group USC (Experimental): Effect of ultrasound cavitation sessions on sex hormones in obese infertile patients with poly cystic ovarian syndrome
  Interventions: Device: Ultrasound cavitation in group A
- Group EA (Experimental): Effect of electro acupuncture on sex hormones in obese infertile patients with poly cystic ovarian syndrome
  Interventions: Device: Electro acupuncture in group B

INTERVENTIONS:
Device: Ultrasound cavitation in group A — Group A:
  twenty obese infertile patients with PCO who will be treated by ultrasound cavitation, 2 times per week for 3 months with medical treatment and hypocaloric diet (1200 kcal/day)
  Arms: Group USC
Device: Electro acupuncture in group B — Group B:
  twenty obese infertile patients with PCO who will be treated by electroacupuncture, 3 times per week for 3 months with medical treatment and hypocaloric diet (1200 kcal/day)
  Arms: Group EA

SUMMARY:
The aim of this study is to determine the difference between the effect of Ultrasound Cavitation and Elctroacupuncture on sex hormones in obese infertile patients with poly cystic ovarian syndrome …………………………………………………………………… BACKGROUND: Polycystic ovary syndrome (PCOS) is a common endocrine and metabolic disorder that occurs in 6 - 10% of women at the reproductive age. It is associated with an-ovulation, infertility, hyperandrogenism, obesity and insulin resistance.

Endocrine characteristics of PCOS are elevated serum concentrations of androgens and Luteinizing hormone (LH) and decreased concentrations of sex hormone binding globulin (SHBG).

Ultrasound cavitation is the method in handling Subcutaneous Adipose Tissue (, especially in destroying subcutaneous fat and shaping a particular part of the body. As one of the non-surgical correction method, UC is preferred for lowering the risk of complications due to obesity.

UC reported a greater decrease of the WHR, suggesting a valuable modification of fat distribution pattern, especially at the abdominal level. It improves rates of ovulation, provides higher incidence of regular menstrual cycles and lower levels of total testosterone.

Acupuncture is a treatment method used in Traditional Chinese Medicine. Electroacupuncture promotes follicle development and corrects reproductive endocrine dysfunction in ovaries by regulating the functions of the hypothalamus, pituitary and ovaries

DETAILED DESCRIPTION:
This study will be designed as prospective, randomized, single blind, experimental, pre-post test , controlled- trial study.

Simple Size Calculation:

I- Subjects:

Forty obese infertile patients with poly cystic ovarian syndrome will participate in this study to determine the difference between the effect of Ultrasound Cavitation and Elctroacupuncture on sex hormones. They will be selected randomly from Out Patient Clinic of Aga Hospital Central, in Aga. All patients will be divided randomly into two equal groups (A&B).

Group A:

twenty obese infertile patients with PCO who will be treated by ultrasound cavitation, 2 times per week for 3 months with medical treatment and hypocaloric diet (1200 kcal/day)

Group B:

twenty obese infertile patients with PCO who will be treated by electroacupuncture, 3 times per week for 3 months with medical treatment and hypocaloric diet (1200 kcal/day) II- Instrumentations:

1. Recording data sheet (Appendix II).
2. Standard weight height scale: measure BMI
3. Tape measurement: measure waist/hip ratio.
4. Test tubes: used to collect the blood samples from obese infertile patients
5. Kites: used for assessment of serum progesterone level, testosterone, LH and FSH.
6. Abdominal ultrasongraphy: measure ovulation rate.
7. cavitation in group A 8- electroacupuncture in group B

ELIGIBILITY:
Inclusion Criteria:

1. Their ages will be ranged between 20-35 year old.
2. Their body mass index will be ranged from 30-40 kg/m2.
3. All of them are married women.

Exclusion Criteria:

* Women will be excluded if they have one of the following criteria:

  1. Diabetes mellitus.
  2. Thyroid dysfunction.
  3. Concomitant cardiovascular disorders.
  4. Respiratory, renal and liver dysfunction.
  5. Tubal adhesions as well as uterine abnormalities.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
weight | up to 12 weeks
  It will be use weight scale to measure weight to calculate the body mass index (BMI) for each woman.
waist/hip ratio: | up to 12 weeks
  It will be use tape measurement to calculate the waist/hip ratio.
Testosterone hormones : | up to 12 weeks
  They will be use kites for assessment of level of testosterone hormones
FSH Hormone | up to 12 weeks
  They will be use kites for assessment of level of FSH hormones
Lh hormones | up to 12 weeks
  They will be use kites for assessment of level of LH hormones
Progesterone hormones | up to 12 weeks
  They will be use kites for assessment of level of progesterone hormones
Height | up to 12 weeks
  It will be use tape measurement to measure height to calculate the body mass index (BMI) for each woman.

SECONDARY OUTCOMES:
Ovulation rate | up to 12 weeks
  It will be use ultrasonography for measuring ovulation rate.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From may 2021 to may 2022

DOCUMENTS (1):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT04875312/Prot_000.pdf